CLINICAL TRIAL: NCT03920735
Title: Retrospective Non-interventional Analysis of Opportunistic Infections in Immunocompromised and Frail Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 1INFOPP
Record Dates: First submitted 2018-08-06; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2018-09

CONDITIONS: Hematologic Disease; Neoplams; Transplantation; Immunologic Deficiency Syndromes; Critical Illness
MeSH Terms: conditions — Hematologic Diseases; Immunologic Deficiency Syndromes; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Opportunistic infection: Immunocompromised or frail patients with an opportunistic infection
- Control group: Immunocompromised or frail patients with no opportunistic infection

SUMMARY:
The analysis of a cohort of consecutive non-selected patients from the Strasbourg University Hospital, and therefore representative of the real life, will allow better identifying the risk factors for these infections (by comparison with a cohort of patient with similar conditions of immunosuppression and no infection) and improving the diagnosis and therapeutic management.

The primary objective is to identify prognosis factors affecting survival in patients with opportunistic infections

ELIGIBILITY:
Inclusion criteria:

* Non selected consecutive immunocompromised or frail patients with an opportunistic infection
* Hospitalized in any of the department of the University Hospital of Strasbourg
* For epidemiological study, patients with similar immunodepression of frail condition and no opportunistic infection

Exclusion criteria:

- Opposition of the patient to use his personal data

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in any department of the University Hospital of Strasbourg since 1997 Opportunistic infectious disease occurrence in immunocompromised or frail patients.
  In case of epidemiological study, patients from a control group with the same characteristics but without infection can be included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
Short- and long-term survival, overall and in specific subgroups of patients | Long-term time point : 1st may 2019
Short- and long-term survival, overall and in specific subgroups of patients | Short term : 1 month
Short- and long-term survival, overall and in specific subgroups of patients | Short term : 3 months
Short- and long-term survival, overall and in specific subgroups of patients | Short term : 6 months

SECONDARY OUTCOMES:
Risk factors predisposing to opportunistic infections - age - gender - Type of work - Location - Tobacco use | first day of opportunistic infection
Prognosis factors in patients with opportunistic infection affecting the response to antimicrobial therapy (using response criteria defined by EORTC/MSG) | first day of opportunistic infection
Identification of baseline prognosis factors affecting the 3 months survival | first day of opportunistic infection
Identification of baseline prognosis factors affecting the 6 months survival | first day of opportunistic infection
Incidence of specific opportunistic infections in different host groups | evolution of a 20-year-period
Description of imaging patterns opportunistic infections: analysis of chest CT-scan and cerebral CT-scan and MRI by radiologists | at first day of infection and up to 12 weeks
Assessment of performance of Aspergillus galactomannan detection test in serum | at onset and up to 1 week
Assessment of performance of Aspergillus galactomannan detection test in bronchoalveolar lavage | at onset and up to 1 week
Response rate | at 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raoul HERBRECHT, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided